CLINICAL TRIAL: NCT03640663
Title: The Palestinian Midwifery-led Continuity Model's Effect on Mothers' and Babies' Health Outcomes
Brief Title: Validation of a Midwifery Model in Palestine 2
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Collaborators: University of Oslo (Other)
Responsible Party: Principal Investigator, Erik Fosse, Professor, Head of Department, Oslo University Hospital
Other Study IDs: Midwif2
Record Dates: First submitted 2018-08-07; First posted 2018-08-21 (Actual); Last update posted 2019-02-28 (Actual); Status verified 2019-02

CONDITIONS: Prenatal Care
Keywords: Midwifery-led continuity of care; Birth complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 9 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Midwife led continuity model of care: Women who received antenatal care from midwives from the hospital reaching out to the rural villages
  Interventions: Other: Midwife led continuity model of care
- Regular care group: Women who received care from doctors, nurses or midwives employed at primary Health care centres in rural villages

INTERVENTIONS:
Other: Midwife led continuity model of care — Midwives from the hospitals provided outreaching caseload ante- and postnatal care to women in rural villages clinics and homes
  Groups: Midwife led continuity model of care

SUMMARY:
A midwife-led continuity model of care was implemented in governmental maternal facilities in Palestine. Midwives from the hospitals provided outreaching caseload ante- and postnatal care to women in rural villages clinics and homes. This study investigated if the model had impact on important maternal and neonatal health outcomes. A retrospective cohort design was used.

DETAILED DESCRIPTION:
Background: A midwife-led continuity model of care was implemented in governmental maternal facilities in Palestine. Midwives from the hospitals provided outreaching caseload ante- and postnatal care to women in rural villages clinics and homes. This study investigated if the model had impact on important maternal and neonatal health outcomes.

Method: A retrospective cohort design was used. Nablus governmental hospital, Rafidia's medical records were reviewed and data extracted involving 2199 women with singleton pregnancies, residing in rural villages, and their new-born babies born between January 2016 and February 2017. Outcomes were limited to the available information in the hospital's birth registry. Important maternal outcomes were postpartum anaemia (Hb <11), mode of delivery and induction of labour. Important outcomes for new-borns were premature delivery < 37 weeks, birth weight < 2500g and 1500g and referral to neonatal intensive care unit. Outcomes were compared between women receiving the midwife-led continuity model of antenatal care and women receiving regular care.

ELIGIBILITY:
Inclusion Criteria:

* Women with singleton pregnancies residing in rural areas giving birth at Nablus governmental hospital, Palestine

Exclusion Criteria:

* Multiple pregnancies
* Women residing in urban areas

Ages: 15 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Pregnant women
Study Population: Palestinian women With singleton pregnancies
Sampling Method: Non-Probability Sample
Enrollment: 2199 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2017-02-28 (Actual); Study Completion 2018-08-30 (Actual)

PRIMARY OUTCOMES:
Emergency Caesarean section rate | 17 months
  Percentage of women undergoing emergency Caesarean section

SECONDARY OUTCOMES:
Premature birth rate | 17 months
  Babies born before 37 weeks gestational age
Post partum anaemia in the mother | 17 months
  Low Hb Level at discharge from hospital
Induction of Labour rate | 17 months
  The rate of women in each group who received induction of labour
Birth weight | 17 months
  Weight immediately post partum: Low (<2500g) Very low (<1500)
APGAR score 5 minutes post partum | 17 months
  APGAR score
Referral to neonatal intensive care | 17 months
  Rate of babies that were referred to neonatal intensive care during hospital stay
Blood transfusion rate post partum | 17 months
  Rate of women receiving blood tranfusion during the hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Erik Fosse, Phd, Principal Investigator — Oslo University Hospital
Locations (1):
- Palestinian Ministry of Health, Nablus, West Bank, Palestinian Territories

IPD SHARING:
Plan to Share IPD: Undecided
IPD can be obtained upon approval of the Palestinian Ministry of Health